CLINICAL TRIAL: NCT05791058
Title: Post-Operative Analgesic Efficacy Of Ultrasound Guided Pericapsular Nerve Group Block Versus Combined Suprascapular And Axillary (Circumflex) Nerve Block For Patients Undergoing Shoulder Arthroscopy: A Randomized Controlled Trial
Brief Title: Post-Operative Analgesic Efficacy Of Ultrasound Guided Pericapsular Nerve Group Block Versus Combined Suprascapular And Axillary (Circumflex) Nerve Block For Patients Undergoing Shoulder Arthroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, Assistant Professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ain Shams university 17
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, General; Nerve Block

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (ultrasound guided pericapsular nerve group shoulder block) (Active Comparator)
  Interventions: Procedure: ultrasound guided pericapsular nerve group shoulder block
- Group B( ultrasound guided suprascapular and axillary nerve block) (Active Comparator)
  Interventions: Procedure: ultrasound guided suprascapular and axillary nerve block
- control group (Active Comparator)
  Interventions: Other: general anesthesia without nerve block

INTERVENTIONS:
Procedure: ultrasound guided pericapsular nerve group shoulder block — The patient's arm is placed in external rotation and abducted at 45 degrees. A linear ultrasound probe will be placed longitudinally between the coracoid and the humeral head. After defining the humeral head, the tendon of the subscapular muscle and the deltoid muscle over it, a 50-mm needle will be inserted using the ''in plane'' technique. When the needle pass through the deltoid muscle and touched the subscapularis tendon, a bone-like hard tissue will be felt and the needle could not be advanced further. The needle tip will be placed between the deltoid muscle and subscapularis tendon, and 20 cc of 0.25% bupivacaine hydrochloride with 4mg dexamesathone will be injected
  Arms: Group A (ultrasound guided pericapsular nerve group shoulder block)
Procedure: ultrasound guided suprascapular and axillary nerve block — The patient will be positioned in a semi-recumbent position with the operating arm on the contralateral shoulder. The probe will be kept over the scapular spine to identify the trapezius and the supraspinatus muscle. Then, it will be moved laterally to identify the concavity of the supraspinatus fossa and the hyper-echoic fascia of the supraspinatus muscle. In the concavity of the fossa, the suprascapular artery and the suprascapular nerve run in close proximity. 10 ml of 0.25% bupivacaine with 2mg dexamethasone will be injected below the supraspinatous fascia then the posterior surface of the humerus will be visualised in the short axis view. So, the AN and posterior circumflex artery will be visualised longitudinally. 10 ml of 0.25% bupivacaine with 2mg dexamethasone will be injected into space
  Arms: Group B( ultrasound guided suprascapular and axillary nerve block)
Other: general anesthesia without nerve block — this group will receive general anesthesia without nerve block
  Arms: control group

SUMMARY:
Recently, the Combined suprascapular nerve block and axillary nerve block (SSNB+ANB) was proposed to provide anesthesia and postoperative analgesia for shoulder surgery as a safe alternative to interscalene block. These two peripheral nerves are responsible for the majority of the sensory innervation of the shoulder.

PENG block has been studied extensively in hip surgeries, but its place in shoulder surgeries is not yet clear. It is a new technology reported for block of articular branches of the shoulder and well pericapsular spread around the glenohumeral joint Therefore, achieving pain relief while avoiding motor block allows us not only to provide an early rehabilitation program in the postoperative period, but also to control the chronic nociceptive activation secondary to pain-induced movement

DETAILED DESCRIPTION:
Preoperative:

Routine preoperative assessment will be done before operation to all patients including history, clinical examination and laboratory investigations (complete blood picture, kidney function tests, liver function tests, pro-thrombin time, and partial thromboplastin time). Chest X-ray, electrocardiogram [ECG] will be done for patients above 40 years old.

All patients will be informed about the study design and objectives as well as tools and techniques. Informed consent will be signed by every patient prior to inclusion in the study.

All patients will be informed about the analgesic regimen and will be instructed on how to express pain intensity with use of the visual analogue scale (VAS) (10cm unmarked line in which 0=no pain, 10cm=the worst imaginable pain)

Anesthetic techniques:

1. General Anesthesia Technique:

   Pre-medications will be given to every patient of the two including groups in the form of midazolam (0.05 mg/kg, IV) together with omeprazole (40 mg, IV) and ondansetron (4 mg, IV) on arrival to the operative room after establishing a peripheral intravenous access. Vital signs will be continuously monitored. After pre-oxygenation for 3 minutes, general anesthesia is induced to all patients with fentanyl (1-2 μg/kg, IV), propofol (1-2mg/Kg, IV), and atracurium (0.5mg/Kg, IV) to facilitate endotracheal intubation. Intermittent positive pressure ventilation of both lungs will be applied (to maintain O2 saturation >98% and end tidal carbon dioxide measurement around 35-38 mmHg). Maintenance of anesthesia will be achieved using intermittent positive pressure ventilation with inhalation of 1-1.5% isoflurane in 50% O2 and atracurium (0.1mg/Kg, IV) every 30 minutes to maintain muscle relaxation.
2. Ultrasound guided PENG shoulder block Technique (Group A):

   The patient's arm is placed in external rotation and abducted at 45 degrees. A linear ultrasound probe will be placed longitudinally between the coracoid and the humeral head. After defining the humeral head, the tendon of the subscapular muscle and the deltoid muscle over it, a 50-mm needle will be inserted using the ''in plane'' technique. When the needle pass through the deltoid muscle and touched the subscapularis tendon, a bone-like hard tissue will be felt and the needle could not be advanced further. The needle tip will be placed between the deltoid muscle and subscapularis tendon, and 20 cc of 0.25% bupivacaine hydrochloride with 4mg dexamesathone will be injected.
3. Ultrasound guided combined suprascapular nerve block and axillary nerve block (SSNB+ANB) Technique (Group B):

The ultrasound guided suprascapular nerve block:

The patient will be positioned in a semi-recumbent position with the operating arm on the contralateral shoulder. The probe will be kept over the scapular spine to identify the trapezius and the supraspinatus muscle. Then, it will be moved laterally to identify the concavity of the supraspinatus fossa and the hyper-echoic fascia of the supraspinatus muscle. In the concavity of the fossa, the suprascapular artery and the suprascapular nerve run in close proximity. 10 ml of 0.25% bupivacaine with 2mg dexamethasone will be injected below the supraspinatus fascia.

The ultrasound guided axillary nerve block:

The patients is positioned in a semi-recumbent position with the arm slightly flexed and adducted at the elbow. The posterior surface of the humerus will be visualised in the short axis view. So, the AN and posterior circumflex artery will be visualised longitudinally. 10 ml of 0.25% bupivacaine with 2mg dexamethasone will be injected into space.

The blocks will be considered a failed block if the block is not successful 30 min after the injection of the local anaesthetic.

Group A 20 Patients of this group will receive ultrasound guided pericapsular nerve group shoulder block (PENG Block) at the end of surgery using 20 ml of 0.25% bupivacaine with 4mg dexamethasone with a maximum dose of (3mg/kg).

Group B 20 Patients of this group will receive single shot suprascapular and axillary nerve using a single dose of 10ml of 0.25% bupivacaine with 2mg dexamethasone each at the end of surgery for postoperative pain relief.

Group C 20 patients of this group will receive general anesthesia without nerve block. In the post anesthesia care unit (PACU) for first hour and in ward afterwards , all patients will be assessed for presence and severity of pain at at 1, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hours postoperatively or at any time patient suffers from pain with visual analog score and recording its value at any patient visit.

Nalbuphine 0.1 mg/kg is the rescue analgesic that will be given to any patient who will suffer pain with VAS more than 3.

ELIGIBILITY:
Inclusion Criteria:

* Adults between age of 18 and 60 years old undergoing elective shoulder arthroscopy surgery.
* American society of anesthesiologists classification (ASA) Ⅰ&Ⅱ
* Males & Females

Exclusion Criteria:

* Age: < 18 or > 60 years old.
* Patients refuse to participate in the study.
* Patients with known hypersensitivity to local anesthetics.
* Coagulation disorder
* Infection at the site of injection
* Hepatic impairment
* Renal impairment
* Severe intraoperative bleeding affecting the hemodynamics status of the patient.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-05-20 (Estimated); Primary Completion 2023-05-20 (Estimated); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
visual analogue score | immediately after extubation
  A scale from 0-10 was allocated with 0 representing no pain and 10 representing the worst imaginable pain
visual analogue score | 2 hours postoperative
  A scale from 0-10 was allocated with 0 representing no pain and 10 representing the worst imaginable pain
visual analogue score | 4 hours postoperative
  A scale from 0-10 was allocated with 0 representing no pain and 10 representing the worst imaginable pain
visual analogue score | 8 hours postoperative
  A scale from 0-10 was allocated with 0 representing no pain and 10 representing the worst imaginable pain
visual analogue score | 12 hours postoperative
  A scale from 0-10 was allocated with 0 representing no pain and 10 representing the worst imaginable pain
visual analogue score | 16 hours postoperative
  A scale from 0-10 was allocated with 0 representing no pain and 10 representing the worst imaginable pain
visual analogue score | 24 hours postoperative
  A scale from 0-10 was allocated with 0 representing no pain and 10 representing the worst imaginable pain
visual analogue score | 36 hours postoperative
  A scale from 0-10 was allocated with 0 representing no pain and 10 representing the worst imaginable pain
visual analogue score | 48 hours postoperative
  A scale from 0-10 was allocated with 0 representing no pain and 10 representing the worst imaginable pain

SECONDARY OUTCOMES:
Time time to first dose of rescue analgesic | during 48 hours after operation
Total dose of analgesic needed | during 48 hours after operation
Complications | during 48 hours after operation
  number of participants developed complications

IPD SHARING:
Plan to Share IPD: No